CLINICAL TRIAL: NCT02596724
Title: TME Neoadjuvant Breast Registry (The NEAT Registry)
Brief Title: TME Neoadjuvant Breast Registry
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Targeted Medical Education (Other)
Responsible Party: Sponsor
Other Study IDs: TMENEO-100
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Breast Cancer; Neoadjuvant therapy for breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Genomic and/or molecular testing of blood or tissue — Genomic and/or molecular testing of blood or tissue

SUMMARY:
Prospective observational registry that links results of the genomic and other molecular testing to treatment response and survival measures in patients who have been diagnosed with breast cancer and who are targeted for neo-adjuvant therapy. Analysis includes how tests impact treatment decisions and outcomes.

DETAILED DESCRIPTION:
Physicians will order tests on patients as part of standard of care; they will report whether test results influenced: selection between standard therapies or a clinical trial; offered insight into mid therapy treatment changes; or helped physicians determine what therapy to offer patients who do not have a complete pathologic response. Patient demographics, diagnosis, type of treatment, surgery and pathologic results will be recorded. Patients will be followed for 5 years. Recurrence and survival data will be recorded.

Participating sites will submit de-identified patient data via electronic case report forms (eCRFs) into a secure study website.

All patients are required to sign an Informed Consent Form. All investigators and staff will have Human Subject Protection Training.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven invasive breast cancer who have started or are scheduled to start neo-adjuvant chemotherapy or endocrine therapy
* Ages 18-90
* Written informed consent

Exclusion Criteria:

* Patients who have had excisional biopsy or axillary dissection
* Patients with confirmed metastatic disease
* Patients who have had recent chemotherapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven invasive breast cancer who have started or are scheduled to start neo-adjuvant chemotherapy or endocrine therapy. Aged 18-90.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Pathologic response and/or endocrine sensitivity | Post surgical treatment--usually within 4 months

SECONDARY OUTCOMES:
Metastasis-free/relapse-free survival in molecular subgroups | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pat Whitworth, M.D., Principal Investigator — Nashville Breast Center; Peter Beitsch, M.D., Principal Investigator — Dallas Surgical Group
Locations (4):
- United States (4):
  - Valley Medical Oncology Consultants, Los Gatos, California
  - Coordinated Health Breast Care Specialists, Allentown, Pennsylvania
  - Nashville Breast Center, Nashville, Tennessee
  - Dallas Surgical Group, Dallas, Texas